CLINICAL TRIAL: NCT05035173
Title: Women's Cancer Survivorship: The LYSA (Linking You to Support and Advice) Trial
Brief Title: The LYSA (Linking You to Support and Advice) Trial
Acronym: LYSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other); Irish Cancer Society (Other); Breakthrough Cancer Research (Unknown); Cancer Research@UCC (Unknown); Cancer Trials Cork (Unknown); Clinical Research Facilites - Cork (CRF-C) (Unknown); Cork University Hospital (Other); Enhancing Cancer Awareness and Survivorship Programmes (ECASP) (Unknown)
Responsible Party: Principal Investigator, Roisin Connolly, Professor, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R19258; WHI19CON (Other Grant/Funding Number: Irish Cancer Society); BCR-2019-09-ICS-UCC (Other Grant/Funding Number: Breakthrough Cancer Research)
Record Dates: First submitted 2021-04-26; First posted 2021-09-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Survivorship; Breast Cancer; Cervical Cancer; Endometrial Cancer
Keywords: Survivorship; Complex Interventional Study; Randomised; Electronic Patient Reported Outcomes; Breast Cancer; Cervical Cancer; Endometrial Cancer; Nurse Lead Clinic; Dietitian Intervention; Nurse intervention; Symptom Management; Quality of Life; Self-care Agency
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Participants will have available the services offered by the Women's Cancer Survivorship Clinic and will undertake electronic Patient Reported Outcomes at baseline, 2, 4, 6, 8, 10, 12 months (end of the study).
  Interventions: Other: Survivorship Clinic Assessments; Other: Survivorship Clinic Nurse Resource; Other: Survivorship Clinic Dietitian Resource
- Control Arm (Active Comparator): Participants will attend a baseline and end of the study visit (12-month time point) to the Women's Cancer Survivorship Clinic to undertake the baseline and complete end of study assessments. They will complete ePRO at baseline and at 12 months. They will have usual follow up care over the 12 month period of the study. Where participants in the control arm contact the Survivorship team for clinical or other advice, they will be referred to the usual care pathway.
  Interventions: Other: Survivorship Clinic Assessments

INTERVENTIONS:
Other: Survivorship Clinic Assessments — Patients will visit in person the Survivorship Clinic at the baseline and end of the study (12-month) at the ORCHID center in the Cork University Hospital (Cork, Ireland).
  During these visits, baseline and end of the study assessments will be made. Patients will receive routine standard information, a care plan and resources about survivorship at the baseline visit.
Other: Survivorship Clinic Nurse Resource — Patients will receive a Survivorship Personal Treatment Plan by the nurse from the Women's Health Initiative Survivorship Clinic according to the results from the baseline ePROs. In addition to that, each 2 months for a period of 12 months, the patient will be answering ePROs. The nurse will undertake an intervention when needed based as per the Trigger system (developed form ePROs responses) or clinical judgement.
  - ePRO Symptom Survey Instrument (nurse questions): A core list of symptoms/adverse events that are identified including gastrointestinal, attention/memory, pain, fatigue and insomnia, mood-emotional distress/depression, anxiety, fear of cancer recurrence, gynaecological, urinary, sexual issues, hot flashes.
  Other Names: Complex Intervention
  Arms: Intervention Arm
Other: Survivorship Clinic Dietitian Resource — Patients will receive Diet Education and Personalised Nutrition Counselling by the dietitian from the Women's Health Initiative Survivorship Clinic at the baseline. In addition to that, each 2 months for a period of 12 months, the patient will be answering ePROs. The dietitian will undertake an intervention when needed as per the Trigger system (developed form ePROs responses) or clinical judgement.
  - ePRO Symptom Survey Instrument (diet questions): nutritional risk (lack of appetite; worry regarding weight loss; worry regarding weight gain), weight, and exercise.
  Other Names: Complex Intervention
  Arms: Intervention Arm

SUMMARY:
This study's aim is to evaluate the feasibility of introducing a women's malignancy survivorship clinic incorporating symptom management through ePRO collection (complex intervention) into routine follow up care in patients with early-stage Hormone Receptor(HR)-positive breast and gynaecologic cancer post primary curative therapy.

DETAILED DESCRIPTION:
Study Design: Complex interventional study. Specific Aims: To evaluate the feasibility of introducing a women's malignancy survivorship clinic in Ireland incorporating symptom management through electronic Patient Reported Outcomes (ePROs) collection (complex intervention) into routine follow-up care in patients with early-stage HR-positive breast and gynecologic cancer post-primary therapy.

Sampling Method: Randomized Control Design (Parallel Arms). Sample Size: 200.

Entry Criteria: Women with early-stage breast/gynecologic cancer within 12 months of completion of primary curative therapy:

* Breast cancer: Stage I-III hormone receptor-positive (defined as estrogen receptor and/or progesterone receptor ≥ 1%) and HER2-negative per ASCO-CAP guidelines on or recommended to commence adjuvant endocrine therapy during the study period.
* Cervical cancer: Stage I to III treated with curative intent.
* Endometrial cancer: treated with curative intent adjuvant radiotherapy +/- chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Women aged > or = 18 years.
2. Ability to read and understand English.
3. Access to internet.
4. Early-stage breast/gynaecologic cancer within 12 months of completion of primary curative therapy:

   * Breast cancer: Stage I-III hormone receptor-positive (defined as estrogen receptor and/or progesterone receptor ≥ 1%) and HER2-negative per ASCO-CAP guidelines on or recommended to commence adjuvant endocrine therapy during the study period.
   * Cervical cancer: Stage I to III treated with curative intent.
   * Endometrial cancer: treated with curative intent adjuvant radiotherapy +/- chemotherapy

Exclusion Criteria:

1. Patients who are not treated with curative intent as above.
2. Patients with premalignant disease.
3. Persons who, in the opinion of the researcher or supervising clinician, are unable to cooperate adequately with the study protocol.
4. Recent (within 12 months) participation in a study/programme involving a lifestyle intervention (e.g diet, exercise, survivorship). Note: Per discretion of PI as to whether may impact the outcome of this study intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled in the clinic. | At the baseline
  Number of patients who were eligible and accepted to participate in the study. This will be recorded in the electronic Case Report Forms (eCRF).
Reasons for not enrolling to the study. | At the baseline
  The reasons for not enrolling will be asked to the patient considering and clusters of option groups will be done.This will be recorded in the electronic Case Report Forms (eCRF).
Reasons for not completing the intervention (drop out). | During the study period (12-month)
  Patients will be contacted to ask about the reasons for not completing the intervention. This will be recorded in the electronic Case Report Forms (eCRF).
Percentage of adherence to the intervention completing ePROs surveys | Baseline, each 2 months till end intervention (12 months)
  Number of enrolled patients who complete the baseline and follow-up ePRO surveys. This will be recorded in the ePROs.
Number of patients who partake in healthcare professional consultations after ePRO data triggers. | Baseline, each 2 months till end intervention (12 months)
  A trigger system with the ePRO measurements has been developed to assess symptoms deterioration that will require that the nurse or Dietitian contact the patient. This will be recorded in the electronic Case Report Forms (eCRF).
Average consultation time in the Womens Survivorship Clinic. | Baseline, each 2 months till end intervention (12 months)
  Time spent by the Nurse, the Dietitian and other Health Care Professionals (HCP) from the Women Survivorship Clinic during consultation will be collected. This will be recorded in the electronic Case Report Forms (eCRF).

SECONDARY OUTCOMES:
Change from Baseline in cancer-related symptoms scores assessed by Patient-Reported Outcomes. | Both arms at the baseline and at the end of the study (12-month); intervention arm month 2, 4, 6, 8, 10
  The cancer-related symptoms items will be assessed by the validated Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) item library and Patient-Reported Outcomes Measurement Information System (PROMIS) item library.
Change from Baseline in Health related-Quality of Life Questionnaire (QLQ) scores assessed by European Organization for the Research and Treatment of Cancer (EORTC). | Both arms at the baseline and at the end of the intervention (12-month)
  All patients will answer at the baseline and at the end of the intervention EORTC QLQ-C30 (30 items). The scoring will be performed according to the EORTC scoring manual. All scores will be linearly transformed to a 0 to 100 scale. A high or healthy level of functioning represents a high functional score.
Change from Baseline in Health related-Quality of Life Questionnaire (QLQ) Breast Cancer Module scores assessed by European Organization for the Research and Treatment of Cancer (EORTC). | Both arms at the baseline and at the end of the intervention (12-month)
  Cohort of patients who had breast cancer will answer at the baseline and at the end of the intervention EORTC QLQ Breast Cancer Module (BR23). The scoring will be performed according to the EORTC scoring manual. All scores will be linearly transformed to a 0 to 100 scale. A high or healthy level of functioning represents a high functional score.
Change from Baseline in Health related-Quality of Life Questionnaire (QLQ) Cervical Cancer Module scores assessed by European Organization for the Research and Treatment of Cancer (EORTC). | Both arms at the baseline and at the end of the intervention (12-month)
  Cohort of patients who had cervical cancer will answer at the baseline and at the end of the intervention EORTC QLQ Cervical Cancer Module (CX24). The scoring will be performed according to the EORTC scoring manual. All scores will be linearly transformed to a 0 to 100 scale. A high or healthy level of functioning represents a high functional score.
Change from Baseline in Health related-Quality of Life Questionnaire (QLQ) Endometrial Cancer Module scores assessed by European Organization for the Research and Treatment of Cancer (EORTC). | Both arms at the baseline and at the end of the intervention (12-month)
  Cohort of patients who had endometrial cancer will answer at the baseline and at the end of the intervention EORTC QLQ Endometrial Cancer Module (EN24). The scoring will be performed according to the EORTC scoring manual. All scores will be linearly transformed to a 0 to 100 scale. A high or healthy level of functioning represents a high functional score.
Change from Baseline in EuroQol 5-Level 5-Dimensions quality-adjusted life-year version (EQ-5D-5L-QALY) scores. | Both arms at the baseline and at the end of the intervention (12-month)
  All patients will answer the EQ-5D-5L-QALY at the baseline and at the end of the intervention. A high score represents high functionality problems.
Change from Baseline in Appraisal Self-Care Agency-R scores (15 items). | Both arms at the baseline and at the end of the intervention (12-month)
  All patients will answer at the baseline and at the end of the intervention the Appraisal Self-Care Agency-R (15 items). The higher the score, the better the self-care agency
Change from Baseline in adjuvant endocrine therapy medication adherence. | Both arms at the baseline and at the end of the study (12-month); intervention arm month 2, 4, 6, 8, 10
  All patients will self-report their adherence at the baseline and at the end of the study. The intervention arm will be asked about it every 2 months.
Assessment of Usability and Satisfaction of the survivorship clinic will be assessed by the Usability and Satisfaction Scale (Lewis, 1995). | Intervention arms at the end of the intervention (12-month)
  Patients in the intervention arm will complete the Usability and Satisfaction Scale (Lewis, 1995) at the end of the intervention. The higher the score, the better usability and satisfaction from the participant.
Experience and opinions from patients, HCP and wider stakeholders about the Women Survivorship Study including the clinic. | Intervention arms at the end of the intervention (12-month)
  Qualitative data collection will be done via Interviews/Focus Groups at the end of the intervention.
Number of resources used by each patient with a cancer related symptom to evaluate the economic impact. | Both arms at the end of the intervention (12-month)
  The main sources from which this data will be collected include: patient hospital record forms, case report forms, use of resources forms, and patient diaries.
Change from Baseline in Diet intake scores from multiple 24-hour recalls, complemented by a Food Frequency Questionnaire (FFQ). | Both arms at the baseline and at the end of the intervention (12-month)
  All patients will answer at the baseline and at the end of the intervention the FFQ. All patients will answer at the baseline and at the end of the intervention the Food Frequency Questionnaire. Data will be entered in to the FFQ European Prospective Investigation into Cancer and Nutrition (EPIC) Tool for Analysis (FETA). FETA calculates the average daily intake of 46 nutrients and 14 food groups, for each individual. The default nutrients list provides a description of each nutrient/food group and the units used. The nutrient data for the FFQ foods have come from McCance and Widdowson's "The Composition of Foods (5th edition)" and its associated supplements.
Change from Baseline in Diet quality scores from The World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) standardised scoring system (Shams-White et al 2019). | Both arms at the baseline and at the end of the intervention (12-month)
  All patients will answer at the baseline and at the end of the intervention the WCRF/AICR. The higher the score, the better Diet quality.
Change from Baseline in BMI scores. | Both arms at the baseline and at the end of the intervention (12-month); intervention arm each 2 months
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. Weight and height will be combined to report BMI in kg/m^2. Patients in the intervention arm will self-report weight in kg every 2 months.
Change from Baseline in Lean Body Mass (LBM) scores. | Both arms at the baseline and at the end of the intervention (12-month)
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. Weight and body fat will be combined to report LBM in kg*(Percentage body/100).
Change from Baseline in waist circumference scores. | Both arms at the baseline and at the end of the intervention (12-month)
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. Waist circumference will be measured in cm.
Change from Baseline in Segmental Body Composition scores assessed measured by Body Composition Monitor bioimpedance spectroscopy (BIS). | Both arms at the baseline and at the end of the intervention (12-month).
  The dietitian will perform physical assessments on each patient at the baseline and at the end of the study. Weight (Kg) and body fat (%) and Total Body Water (TBW) will be combined to report the Body Composition score.
Change from Baseline in muscle strength scores on handgrip measurements. | Both arms at the baseline and at the end of the intervention (12-month)
  The dietitian will perform physical assessments to each patient at the baseline and at the end of the study. Muscle strength will be measured using hand grip strength (HGS) based on the Jamar Dynamometer (Model 091011725).
Change from Baseline in Nutritional risk scores assessed by the Malnutrition Screening Tool (MST). The higher the score, the higher risk of malnutrition. | Both arms at the baseline and at the end of the intervention (12-month)
  All patients will complete the MST at the baseline and at the end of the intervention. Patients in the intervention arm answer the MST each 2 months. The higher the score, the higher risk of malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Kate O Connell, Ms., Study Chair — Research Support Officer Clinical (Nurse Manager); Laia Raigal, Dr., Study Chair — Data Manager
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No
Not applicable at the moment.

REFERENCES:
- [Derived] Kearns N, Raigal-Aran L, O'Connell K, Davis A, Bermingham K, O'Reilly S, Collins DC, Corrigan M, Coulter J, Cleary V, Cushen S, Flavin A, Byrne F, O'Grady A, O'Neill D, Murphy A, Dahly D, Palmer B, Connolly RM, Hegarty J. The Women's Health Initiative cancer survivorship clinic incorporating electronic patient-reported outcomes: a study protocol for the Linking You to Support and Advice (LYSA) randomized controlled trial. Pilot Feasibility Stud. 2022 Nov 10;8(1):238. doi: 10.1186/s40814-022-01186-x. PMID 36357934
- See also: Women's Health Initiative - Cancer survivorship support for women — https://www.cancer.ie/cancer-research/about-our-cancer-research/our-cancer-research-networks/womens-health-initiative
- See also: Women's Cancer Survivorship: Supporting And Innovating For Change — https://www.breakthroughcancerresearch.ie/research/womens-cancer-survivorship/
- See also: Short video about the Women's Health Initiative pilot clinic in Cork — https://www.youtube.com/watch?v=iD5Zdxfm14A